CLINICAL TRIAL: NCT05642676
Title: Welcoming by Design Pilot: Reducing Structural Stigma by Changing Clinic Systems and Architectural Design to Make HIV Clinics More Friendly, Private, and Patient-Centric
Brief Title: Welcoming by Design Pilot: Reducing Structural Stigma by Changing Clinic Systems and Architectural Design
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to obtain funding
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MED-2023-32453'
Record Dates: First submitted 2022-11-08; First posted 2022-12-08 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventions clinics to be remodeled (Experimental)
  Interventions: Other: Clinics remodeling

INTERVENTIONS:
Other: Clinics remodeling — changes to the clinics will be planned based on baseline surveys

SUMMARY:
The purpose of this study is to test the feasibility and acceptability of implementing clinic system changes and physical structures in Uganda to improve aesthetics, welcome, and privacy to reduce HIV stigma, improve retention-in-care, and improve the patient experience.

To evaluate pilot/implementation outcomes, the outcomes of fidelity, feasibility, and acceptability will be assessed prior to intervention. After the changes are done to two HIV interventions clinics, the outcome surveys will assess if the changes were disruptive or impeded the workings of the clinics.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 and older
* Enrolled in the HIV clinics where we are working
* Able to independently consent for interview, survey, or focus group.

Exclusion Criteria:

* Unable to provide consent
* Does not speak English or Luganda (local language around Kampala and Entebbe)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability survey | Baseline
  How well an intervention will be received by the target population and the extent to which the intervention meets the needs of the target population and organizational setting. This will be assessed through qualitative evaluation and a quantitative survey from patients and staff.
Feasibility | baseline
  An assessment of the practicality of a proposed idea or project, by assessing recruitment capacity, and ability to complete proposed modifications in clinics. The intervention will be judged feasible if enrollment and metrics can be completed.
Fidelity to the Intervention | 6-months post intervention
  Assesses whether the intervention was delivered as intended, using the intervention plan/checklist
Outcomes survey | 6-months post intervention
  assesses if the changes were disruptive or impeded the workings of the clinics.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No